CLINICAL TRIAL: NCT02668913
Title: LCC-CARIS-01: A Pilot Feasibility Study to Assess the Use of Molecular Profiling to Determine Choice of Treatment for Patients With Gynecological Cancer
Brief Title: LCC-CARIS-01: Molecular Profiling in Gynaecological Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geoff Hall (Other)
Collaborators: National Health Service, United Kingdom (Other Government)
Responsible Party: Sponsor-Investigator, Geoff Hall, Lead Clinical Investigator, University of Leeds
Organization: University of Leeds (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MO15/302; 15/YH/0493 (Other: Yorkshire & Humber Ethics Committee)
Record Dates: First submitted 2016-01-21; First posted 2016-01-29 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Epithelial Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer; Gynaecological Malignancy
Keywords: gynaecology; Oncology
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic Analysis (Experimental): This arm will be subject to Caris Molecular profiling.
  Interventions: Other: Diagnostic analysis

INTERVENTIONS:
Other: Diagnostic analysis — Molecular profiling

SUMMARY:
This is a pilot feasibility study assessing the use of a commercial molecular profiling service in the UK's National Health Service (NHS). The impact of knowledge of a patient's molecular profile, and the time it takes to generate this knowledge, will be assessed by analysis of changes in physicians' treatment decisions prior to and following generation of a patient's molecular profile. Implications for benefit with therapies recommended by the profile will also be assessed and the following treatment outcomes collected: best response (based on routine clinical, radiological and biochemical assessment), progression free survival ratio (post Caris Molecular profiling versus prior treatment) and overall survival.

DETAILED DESCRIPTION:
The concept of molecular profiling leading to personalised medicine is based on the hypothesis that using treatments selected by a molecular profiling approach favourably changes the clinical course for an individual patient. In order to best determine the next steps in a particular patient's clinical course, it is necessary to understand not only how that patient has been diagnosed, treated and responded to treatment in the past, but also to fully characterize the molecular profile of the patient's tumour, so that the maximum information on potential positive and negative treatment outcome can be gathered.

In this pilot feasibility study, the treatment plans devised for individual patients by their treating oncologists will be assessed. The primary endpoint is the frequency at which the oncologist changes a treatment plan based on the tumour's molecular phenotype and the respective drugs considered to be associated with higher likelihood of benefit or lack of benefit. Ultimately however, the treatment decision remains in the hands of the treating physicians and the study protocol does not prescribe or dictate the use of any particular treatment.

In patients with recurrent ovarian cancer or other gynecological malignancies in which no standard of care is defined, treatments are currently chosen empirically based on population-based response rates. With the use of molecular profiling treating physicians will get a chance to revise their treatment plans and consider the individual molecular profile of each patient's tumour in light of the known predictive power of biomarkers for the efficacy of certain drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent epithelial ovarian, primary peritoneal or fallopian tube cancer OR patients with other gynaecological malignancy in whom the treating physician has made a decision to commence further systemic treatment with hormones or cytotoxic chemotherapy.
* Patient must be fit and willing to receive further treatment
* Plan to commence chemotherapy within 4 weeks of trial entry.
* Adequate tumour tissue, obtained within 36 months of study, must be available for molecular profiling.
* Age ≥ 18 years
* Patients who have fully understood the information provided and who have provided written informed consent.
* Patients for whom relevant pathology specimens are held by Leeds Teaching Hospitals Trust.

Exclusion Criteria:

* Patients receiving treatment as part of a therapeutic trial in which physicians are not able to select any appropriate treatment option.
* Patients who lack capacity to consent to study participation.
* Patients with symptoms that mean it is clinically inappropriate to delay treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
To measure the number of treatment decisions that will be altered by the results of of the Caris molecular profiling report. | 21 days

SECONDARY OUTCOMES:
To analyse best response marker following CMI directed therapy | 3 years
Determine time to treatment failure (TTTF) (defined as the time from completion of prior therapy to start of next treatment) following CMI directed therapy. | 3 years
Study overall survival following CMI directed therapy. | 3 years
Compare the ratio of TTTF after CMI guided therapy to TTTF under previous treatment. | 3 years
Assess cost of treatment with CMI versus originally planned treatment. | 3 years
To analyse quality adjusted life years (QALYs) in patients treated with CMI-directed therapy. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Hall, PhD FRCP, Principal Investigator — University of Leeds
Locations (1):
- Leeds Cancer Centre, Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom